CLINICAL TRIAL: NCT07396571
Title: Development of a Predictive Infection Score in Patients With Hematological Malignancies Colonized by Multidrug-resistant Enterobacteriaceae
Brief Title: Predictive Score in Patients With Hematological Malignancies Colonized by Multidrug-resistant Enterobacteriaceae
Acronym: SCREEN-IN
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: SCREEN-IN
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hemato-oncologic Patients; Colonization; Neutropenia; Enterobacteria Non Susceptible to Carbapenem Carrier; ESBL-producing Enterobacteriaceae Infections
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbiological isolates will be frozen and forwarded to the coordinating centre for Whole Genome Sequencing (WGS). These isolates shall be stored for a maximum period of 25 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this observational study are to identify risk factors for ESBL-producing Enterobacterales and carbapenemase-producing Enterobacterales (CPE) colonization in oncohematological patients with severe neutropenia, and to develop and validate a predictive model of infection caused by ESBL-producing Enterobacterales and CPE in patients previously colonized by the same bacteria.

The main questions the study aims to answer are:

* What are the risk factors for ESBL-producing Enterobacterales and CPE colonization in patients with severe neutropenia?
* Can a predictive model be developed to accurately predict infections in the colonized patients?

Study Design & Participants: Participants will be screened after receiving neutropenia-inducing treatment (e.g., chemotherapy, chimeric antigen receptor T-cell (CAR-T) therapy, or others). A baseline rectal swab will be collected to assess initial colonization status, followed by weekly swabs throughout the duration of neutropenia. Patients will be followed for 120 days from initial screening, during which the study team will record any infections, with an additional 30-day follow-up period. All hospitalization data will be recorded.

DETAILED DESCRIPTION:
An exploratory metagenomics sub-study will be conducted within the study. Its goal is to describe the intestinal microbiome in patients and analyze any correlation between the microbiome and infection and mortality. For logistical reasons, this sub-study will be performed only on patients in the Seville area. This analysis will be performed via sequencing of the 16S ribosomal ribonucleic acid (rRNA) gene.

ELIGIBILITY:
Inclusion criteria

* Patients admitted to Hematology departments with hematological diseases, including: myelodysplastic syndrome, acute myeloid leukemia, acute lymphoblastic leukemia, multiple myeloma, chronic lymphocytic leukemia, chronic myeloproliferative leukemias, lymphomas, or other hematological disorders.
* Patients scheduled to receive treatment for their underlying hematological disease, including myeloablative/cytotoxic chemotherapy, conditioning chemotherapy for hematopoietic stem cell transplantation (autologous, allogeneic, or other types), lymphodepleting chemotherapy for CAR-T cell therapy, and/or other treatments expected to induce neutropenia.
* Patients expected to develop neutropenia (neutrophil count < 0.5 \times 10^9/L, or < 1.0 \times 10^9/L when predicted to fall below 0.5 \times 10^9/L within the next 48 hours) in the coming days.
* Those who have signed the informed consent form.
* Participation in another study is permitted, provided it is observational and does not influence the potential colonization status.

Exclusion criteria

* Psychiatric disorder or inability to understand or follow the protocol instructions.
* Terminally ill patients or those with an estimated life expectancy of less than 30 days.
* Previous enrollment in the study.
* Known prior colonization by ESBL-producing Enterobacteriaceae (ESBL-E) or carbapenemase-producing Enterobacteriaceae (CPE).
* Physician's discretion: The patient's attending physician prefers not to include the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematological diseases, including: myelodysplastic syndrome, acute myeloid leukemia, acute lymphoblastic leukemia, multiple myeloma, chronic lymphocytic leukemia, chronic myeloproliferative leukemias, lymphomas, or other hematological disorders.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
ESBL-producing Enterobacterales and Carbapenem-resistant Enterobacterales (CRE) colonization in oncohematological patients detected by rectal swab | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  A weekly control of colonizations status will be performed via rectal swabs, while the patient is hospitalized.
Neutropenic fever (NF) and/or clinically relevant infection caused by ESBL-producing Enterobacterales and CPE | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  Due to the observational nature of the study, all cases of NF or infection will be registered in the electronic case report form (eCRF)

SECONDARY OUTCOMES:
All cause mortality at 30 and 120 days | 120 day follow-up since inclusion
  Mortality at 30-days after inclusion and mortality at 120-days after inclusion
In case of infection, mortality related to the infection at day 30 and/or recurrence of infection until day 120 | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  For patients with an infection episode, mortality related to the infection and recurrence will be assessed at day 30 of the security follow-up
Length of hospitalisation(s) (in days) | 120 days follow up since inclusion
  Total number of hospitalisation days during the 120 day follow-up.
Data collection on antibiotic usage in Days of treatment (DOT) | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  Data collection on antibiotic usage in days of treatment
Adjustment of empirical or targeted treatment for infections with a confirmed etiological diagnosis | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  Data collection of antibiotic treatment changes from empirical to targeted based on microbiological results.
C. difficile infection | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  Rate of patients presenting confirmed Clostridioses difficile toxin presence
Fungal infection caused by yeast or mold | 120 days follow-up. In case of infection a security follow-up of 30 days will be performed
  Proven, probable or possible fungal infection confirmed by growth of specimen in culture or fungal biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Zaira R. Palacios Baena, MD/PhD, Principal Investigator — Virgen Macarena hospital
Locations (15):
- Spain (15):
  - Hospital Universitario Torrecárdenas, Almería, Andalusia
  - Hospital Universitario De Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario de Vigo, Vigo, Galicia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Virgen de las Nieves Ruiz de Alda, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville

IPD SHARING:
Plan to Share IPD: No